CLINICAL TRIAL: NCT02757404
Title: Impact of Injection Techniques on the Effectiveness of Botulinum Toxin for the Treatment of Post Stroke Upper Limb Spasticity
Brief Title: Meditoxin® Treatment in Patients With Post Stroke Upper Limb Spasticity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MT_PRT_ST04
Record Dates: First submitted 2016-04-25; First posted 2016-05-02 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Muscle Spasticity
Keywords: botulinum toxin; spasticity; injection technique; neuronox; meditoxin
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasonography guidance (Experimental): Ultrasonography guidance injection of Meditoxin®.
  Interventions: Drug: Ultrasonography guidance injection of Meditoxin®.
- Electrical stimulation guidance (Experimental): Electrical stimulation guidance injection of Meditoxin®.
  Interventions: Drug: Electrical stimulation guidance injection of Meditoxin®.
- Manual needle placement (Experimental): Manual needle placement injection of Meditoxin®.
  Interventions: Drug: Manual needle placement injection of Meditoxin®.

INTERVENTIONS:
Drug: Ultrasonography guidance injection of Meditoxin®. — Meditoxin® will be injected to upper limb spasticity by using the ultrasonography guidance.
  Arms: Ultrasonography guidance
Drug: Electrical stimulation guidance injection of Meditoxin®. — Meditoxin® will be injected to upper limb spasticity by using the electrical stimulation guidance.
  Arms: Electrical stimulation guidance
Drug: Manual needle placement injection of Meditoxin®. — Meditoxin® will be injected to upper limb spasticity by using the manual needle placement.
  Arms: Manual needle placement

SUMMARY:
Botulinum Toxin for the Treatment of Post Stroke Upper Limb Spasticity.

DETAILED DESCRIPTION:
This study is "A Multicenter, Prospective, Randomized, Evaluator Blinded, Comparing Phase 4 Study to Evaluate the Impact of Injection Techniques on the Effectiveness of Botulinum Toxin for the Treatment of Post Stroke Upper Limb Spasticity".

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged over 20.
2. Subjects who has grade 1 + and more spasticity at least one of upper limb muscles as measured on Modified Ashworth Scale after stroke.
3. Subjects who was diagnosed stroke at least 1 month prior to study participation.
4. Subjects or legal representatives who voluntarily decided the participation of the study and signed the informed consent.

Exclusion Criteria:

1. Subjects who had spinal injuries to be a factor of spasticity except for stroke prior to study enrollment.
2. Subjects with allergy or hypersensitivity to the Botulinum Toxin.
3. Subjects who have changed the muscle relaxant taking for treatment within past 4 weeks prior to study participation.
4. Subjects who have taken injection treatments using alcohol or phenol in upper limb within past 6 months prior to study participation.
5. Subjects with general neuromuscular synaptic disorder(e.g. Myasthenia gravis, Lambert-Eaton syndrome, Amyotrophic lateral sclerosis).
6. Subjects who have been injected with botulinum toxin within past 3 months before the injection.
7. Subjects who are pregnant or lactating of disagreed to avoid pregnancy during 3 months study period.
8. Subjects who are scheduled to take part in other clinical trial during the study period.
9. Patients who are not eligible for this study at the medical discretion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2016-08-16 (Actual); Study Completion 2016-08-16 (Actual)

PRIMARY OUTCOMES:
Comparison evaluation on improvement rate of spasticity assessed by Modified Ashworth Scale between 3 arms. | 4 weeks

SECONDARY OUTCOMES:
Comparison evaluation on improvement rate of spasticity assessed by Modified Tardieu Scale between 3 arms. | 4 weeks
Comparison evaluation on improvement rate of range of motion on each joint between 3 arms. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MyungEun Chung, Principal Investigator — St. Paul's Hospital, The Catholic University of Korea

IPD SHARING:
Plan to Share IPD: Undecided